CLINICAL TRIAL: NCT07305636
Title: Assessing the Utility of AI Models in MAFLD Diagnosis: Comparison With Traditional Non-Invasive Fibrosis Scores.
Brief Title: AI Models vs Non-Invasive Fibrosis Scores in MAFLD Diagnosis
Acronym: MAFLD-AI
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nahla Ahmed Khalaf, Lecturer of Tropical Medicine and Infectious diseases, Tanta University
Other Study IDs: TANTAU-MAFLD-AI-2025-01
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: MAFLD; AI (Artificial Intelligence)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the accuracy of artificial intelligence (AI) models using FibroScan and clinical data to predict hepatic fibrosis in Egyptian patients with metabolic-associated fatty liver disease (MAFLD). The performance of the AI models will be compared with conventional noninvasive fibrosis scores (FIB-4, APRI, NAFLD fibrosis score, and FAST). The goal is to improve early, noninvasive diagnosis of fibrosis and reduce reliance on liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

- Adults ≥18 years.

Diagnosed with MAFLD according to international criteria (hepatic steatosis with metabolic dysfunction).

Valid FibroScan evaluation with available LSM and CAP values.

Exclusion Criteria:

* Excessive alcohol intake (>30 g/day for men, >20 g/day for women).

Chronic viral hepatitis (HBV or HCV).

Autoimmune hepatitis.

Known malignancy.

Pregnancy.

Refusal to participate.

Min Age: 18 Days | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult Egyptian patients (≥18 years) diagnosed with metabolic associated fatty liver disease (MAFLD) according to international criteria, recruited from the outpatient clinic and FibroScan unit of the Tropical Medicine Department, Faculty of Medicine, Tanta University.
Sampling Method: Non-Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Measure diagnostic accuracy of AI models in predicting hepatic fibrosis stage (F0-F4) | At enrollment (single cross-sectional assessment).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tanta, Egypt